CLINICAL TRIAL: NCT07336303
Title: Comparative Study on the Effect of Auriculotherapy in the Treatment of Postoperative Pain in Outpatient Surgery: Rhizarthrosis. PARALLEL COMPARATIVE STUDY, RANDOMIZED AND DOUBLE-BLIND
Brief Title: Comparative Study on the Effect of Auriculotherapy in the Treatment of Postoperative Pain in Outpatient Surgery: Rhizarthrosis.
Acronym: AURDO II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Bizet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2025-A02330-49
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Pain Following Outpatient Prosthetic Surgery for Rhizarthrosis

STUDY DESIGN:
Intervention Model Description: * Group A (Experimental): Real auriculotherapy + standard medical care
  * Group B (Control): Sham auriculotherapy + standard medical care
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real auriculotherapy + standard medical care group A (Experimental): real auriculotherapy : patients will have a preoperative session carried out within 72 hours before the surgery
  Interventions: Procedure: outpatient prosthetic surgery for rhizarthrosis.
- sham auriculotherapy + standard medical care group B (Sham Comparator): sham auriculotherapy : patients will have a preoperative session carried out within 72 hours before the surgery
  Interventions: Procedure: outpatient prosthetic surgery for rhizarthrosis.

INTERVENTIONS:
Procedure: outpatient prosthetic surgery for rhizarthrosis. — surgery / procedures : Outpatient surgery (thumb osteoarthritis). On the day of the procedure, the patient arrives on an outpatient basis, is positioned on a stretcher, and is then taken to the pre-anesthesia room where regional anesthesia is performed. The block is carried out under ultrasound guidance following a standardized protocol.
  The patient is then transferred to the operating room, where the tourniquet is applied. The surgical technique is endoscopic, following the AGEE method. At the end of the procedure, the surgeon places two or three absorbable sutures (4/0 or 5/0) on the thinnest areas of skin. The sutures are then covered with a dressing.

SUMMARY:
Auriculotherapy has demonstrated promising potential in the management of postoperative pain. Additionally, one study reported encouraging outcomes regarding the reduction of anxiety levels among patients in primary healthcare settings. Nevertheless, further high-quality research is required to substantiate these findings and to support the integration of auriculotherapy into standardized therapeutic protocols.

The objective of this prospective, comparative, double-blind study is to assess the efficacy of auricular acupuncture in the management of postoperative pain following outpatient prosthetic surgery for rhizarthrosis

ELIGIBILITY:
Inclusion Criteria:

* Subject aged over 18 years
* Patients hospitalized for endoscopic treatment of thumb carpometacarpal osteoarthritis (rhizarthrosis)
* Patient with no prior history of auriculotherapy sessions
* No participation in another clinical study
* Subject affiliated with, or beneficiary of, a social security system
* Agrees to complete all study questionnaires

Exclusion Criteria:

* Patient under 18 years of age
* Unable to comply with medical follow-up required for the study
* Adult subject under legal protection, guardianship, or trusteeship
* Patient with neuropathic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain reduction using the Numerical Rating Scale (NRS) questionnaire during the postoperative period from Day 1 to Day 3. From Day 1 to Day 3, Based on Real or Sham Auriculotherapy Sessions | Day 1 to Day 3
  The Numerical Rating Scale (NRS) is a validated, unidimensional tool used to assess pain intensity. Patients are asked to rate their pain by selecting a number that best reflects its severity.
  Valeur minimale :
  0 - corresponds to "no pain".
  Valeur maximale :
  10 - corresponds to "the worst pain imaginable".
  Interprétation générale :
  0 : No pain
  1-3 : Mild pain
  4-6 : Moderate pain
  7-10 : Severe pain

SECONDARY OUTCOMES:
Assessment of the onset of neuropathic pain using the DN4 questionnaire during follow-up. | At baseline and at one-month postoperative follow-up
  The DN4 questionnaire is a validated diagnostic instrument designed to differentiate neuropathic pain from nociceptive pain. It comprises 10 items, including 7 symptom-based descriptors (e.g., burning, painful cold, electric shocks, tingling, pins and needles, numbness, itching) and 3 clinical examination findings (hypoesthesia to touch, hypoesthesia to pinprick, and pain provoked by brushing).
  Minimum score:
  0, indicating the absence of neuropathic pain features.
  Maximum score:
  10, indicating the presence of all evaluated neuropathic characteristics.
  Interpretation:
  A score ≥ 4 is considered the diagnostic threshold and is associated with a high probability of neuropathic pain, based on the tool's validated sensitivity and specificity. Scores < 4 suggest that neuropathic pain is unlikely.
Assessment of analgesic consumption (number, name, and analgesic step) from the end of the hand regional anesthesia until Day 3, and again at one month | from the end of the hand regional anesthesia until Day 3, and again at one month postoperative follow-up
  analgesic consumption (number, name, and analgesic step)
Assessment of patient satisfaction using the CGI-C scale. | at one-month postoperative follow-up
  The CGI-C is a validated clinician-rated scale used to assess the patient's overall change in clinical status compared with baseline. It provides a global, integrative judgment that incorporates all available clinical information, including symptoms, functioning, and therapeutic response.
  Minimum score: 1 - Very much improved
  Maximum score: 7 - Very much worse
  Interpretation:
  1-2: Marked or clear improvement
  3: Minimal improvement
  4: No change
  5: Minimal worsening
  6-7: Clear to marked worsening
Assessment of postoperative anxiety reduction between the two groups using the State-Trait Anxiety Inventory (STAI) score. | At baseline and at one-month postoperative follow-up
  State-Trait Anxiety Inventory (STAI - Form Y)
  The State-Trait Anxiety Inventory is a validated psychometric instrument designed to assess two distinct components of anxiety:
  State Anxiety (STAI-S): reflects a transient emotional condition characterized by feelings of tension, apprehension, and heightened autonomic activity. It measures anxiety "right now, at this moment."
  Trait Anxiety (STAI-T): reflects a stable predisposition to perceive situations as threatening and to respond with elevated anxiety across time.
  Each subscale contains 20 items, rated on a 4-point Likert scale.
  * Minimum score: 20
  * Maximum score: 80
  Interpretation:
  Higher scores indicate higher levels of anxiety.
  * 20-37: low anxiety
  * 38-44: moderate anxiety
  * ≥ 45: high anxiety

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Benkessou, Paris
  - Bizet Clinic, Paris

IPD SHARING:
Plan to Share IPD: Undecided